CLINICAL TRIAL: NCT05196347
Title: Efficacy and Safety of Dapagliflozin in Patients with Chronic Kidney Disease Stage 4-5 Under Integrated CKD Care Program: an Investigator-led, Randomized, Open-label, Blinded-endpoint, Multicenter Study
Brief Title: Dapagliflozin and Renal Surrogate Outcomes in Advanced Chronic Kidney Disease
Acronym: DAPA-advKD
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Kaohsiung Medical University (Other)
Responsible Party: Principal Investigator, Chi-Chih Hung, Professor, Kaohsiung Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ESR-21-21200 V1.4
Record Dates: First submitted 2021-12-21; First posted 2022-01-19 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2025-03

CONDITIONS: Chronic Kidney Diseases
MeSH Terms: conditions — Renal Insufficiency, Chronic | interventions — dapagliflozin

STUDY DESIGN:
Intervention Model Description: To determine if dapagliflozin + integrated CKD care program is more effective in reducing renal function progression than integrated CKD care program
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- dapagliflozin + integrated CKD care program (Experimental): Subjects will be received dapagliflozin 5 mg for 4 weeks. Uptitration to 10 mg will be done between 5 to 12th weeks, if eGFR dip <20%.
  In both arms, the integrated CKD care program includes CKD stage 4 and 5 education, diet counseling, bioimpedance and echocardiography measurements to control overhydration at 0-1 liter (by body composition monitor (BCM; Fresenius))
  Interventions: Drug: Dapagliflozin
- integrated CKD care program (Active Comparator): In both arms, the integrated CKD care program includes CKD stage 4 and 5 education, diet counseling, bioimpedance and echocardiography measurements to control overhydration at 0-1 liter (by body composition monitor (BCM; Fresenius))
  Interventions: Drug: Dapagliflozin

INTERVENTIONS:
Drug: Dapagliflozin — In dapagliflozin arm, subjects will be received dapagliflozin 5 mg for 4 weeks. Uptitration to 10 mg will be done between 5 to 12th weeks, if eGFR dip <20%.
  Other Names: Integrated CKD care program

SUMMARY:
This is an investigator-led, randomized, open-label, blinded-endpoint, multicenter study that will include a total of approximately 180 subjects from 2 sites. Subjects with an estimated glomerular filtration rate (eGFR) of 10 to 30 mL/min/1.73m2 will be included. The goal of this study is to assess the efficacy and safety of dapagliflozin (Forxiga®, AstraZeneca) in reducing renal function progression and complications of chronic kidney disease (CKD) in patients with CKD stage 4 and 5 under the integrated CKD care. Subjects will be allocated to integrated CKD care program + dapagliflozin or integrated CKD care program alone. The primary endpoint is eGFR decline after randomization between 2 arms. The secondary endpoints are renal and cardiovascular composite outcomes.

DETAILED DESCRIPTION:
eGFR 30 mL/min/1.73m2 is a clinical cut point, below which advanced chronic kidney disease (CKD) (stage 4 and 5) is associated with a significantly increased risk of mortality and a 50-fold increased requirement of renal replacement therapy (RRT). Physicians are suggested to refer patients to nephrologists when eGFR <30 mL/min/1.73m2 for multidisciplinary care. The pre-ESRD care program of CKD stage 3b-5 patients in Taiwan for modifiable risk factors of CKD progression and for preparation of renal replacement therapy (RRT) has shown to improve clinical outcomes.

"Advanced" CKD was usually viewed as "predialysis" CKD and sometimes used interchangeably, probably because of limited time of treatment and limited medications in advanced CKD. The time of treatment in CKD stage 4 in our cohort (median survival of RRT or mortality) was still up to 4.7 (IQR 2.1-8.7) years under the practice of late dialysis initiation (median eGFR 5 mL/min/1.73m2). However, renin-angiotensin system blockade was the only effective medication in patients with advanced CKD, implied by albuminuria reduction and proved for reduction of renal outcome only in some randomized controlled trials (RCTs). Furthermore, there is no effective medication for patients with normoalbuminuria, tubulointerstitial nephropathy, hyperkalemia or blood pressure <130/80 mmHg. Thus, the unmet need in advanced CKD patients is the lack of effective medication.

Recently, two large renal outcome RCTs of sodium-glucose co-transporter 2 inhibitors (SGLT2is), which has been developed as an oral anti-hyperglycemic agent for type 2 diabetes mellitus (T2DM), show a reduction of renal composite outcome and probably of mortality in CKD stage 2 and 3 (CREDENCE and DAPA-CKD trials). Subgroup analyses show similar reduction of renal composite outcome in patients with or without diabetes, albuminuria, or high blood pressure. Consistent with previous large cardiovascular (CV) outcome trials, patients with eGFR 25-30 mL/min/1.73m2 also suggest promising benefits.

Beside, in view of the high atherosclerotic CV risk in advanced CKD, SGLT2is show a reduction of major adverse cardiovascular event in large CV outcome RCTs in T2DM, especially in patients with high CV risk. Also considering the high incidence of cardiorenal syndrome and fluid overload in advanced CKD, SGLT2is show a reduction of congestive heart failure (CHF) event in large CHF RCTs, regardless of T2DM and regardless of preserved or reduced ejection fraction. Analysis in patients with eGFR <30 mL/min/1.73m2 suggest similar protection for atherosclerotic and CHF events.

Diuresis is an important mechanism of the benefit of SGLT2i as observed in the above renal and CV RCTs. Our previous studies demonstrated that overhydration measured by bioimpedance is associated with renal function progression and all-cause mortality. SGLT2i improves overhydration in studies. We would further ask whether the cardiorenal effect of SGLT2i is independent of its diuretic effects in advanced CKD patients.

Study in advanced CKD is difficult. In theory, SGLT2i could decrease hyperfiltration in the residual glomeruli in advanced CKD. Our preliminary data showed some improvements in certain types of advanced CKD after SGLT2i treatment. However, a "Point of no return" theory suggests medication may not alter the natural history of progressive deterioration in renal function in advanced CKD. Subjects with advanced CKD may be at higher risk of adverse effects of the medication being tested. Overall, our integrated CKD care program based on the KDIGO 2017 conference on the prognosis of CKD stage 4 and 5, which emphasizes on the monitoring of diet, blood pressure, fluid status and cardiac function, could be the foundation of treatment in advanced CKD.

Thus, the goal of this study is to assess the efficacy and safety of dapagliflozin (Forxiga®, AstraZeneca) in reducing renal function progression and complications of CKD in patients with CKD stage 4 and 5 under the integrated CKD care and to find out the target subgroups for future RCT.

Study design This is an investigator-led, randomized, open-label, blinded-endpoint, multicenter study that will include a total of approximately 180 subjects from 2 sites. The study design is shown in Figure 1. Subjects with an eGFR of 10 to 30 mL/min/1.73m2 within the 6 months prior to screening will be eligible for screening. Subjects must have at least 3 eGFR measurements in previous 1 year and at least 9 months between first and last eGFR measurements to calculate eGFR decline. Subjects must be in the pre-ESRD care and education program of Ministry of Health and Welfare of Taiwan for 1 month with stable renin-angiotensin system blockade, anti-hypertensive, diuretics and anti-hyperglycemic therapy. In the 4-week screening phase, review of medical history, renal echography, cardiac echography and bioimpedance analysis will be done to assure the safety of study drug treatment. Education for self-monitoring of blood pressure and blood sugar (in diabetes) will also be done.

Qualified subjects will enter the study phase at the randomization visit and will be randomized 2:1 to either integrated CKD care program + dapagliflozin or integrated CKD care program. In both arms, the integrated CKD care program, including CKD stage 4 and 5 education, diet counseling, fluid status and cardiovascular measurements, which is more intensive than the pre-ESRD program, will be done as scheduled in table 1 to control relative overhydration <15% by bioimpedance spectroscopy (BCM; Fresenius). In dapagliflozin arm, subjects will be received dapagliflozin 5 mg for 4 weeks. Uptitration to 10 mg will be done between 5 to 12th weeks, if eGFR dip <20%. Education for drug safety of dapagliflozin will be done.

Subjects will return to the clinic for 4 times in the first 24 weeks (intensive monitor) and return to the clinic every 12 weeks thereafter (regular monitor). Laboratory assessments, measurements, concomitant medication review, adverse event collection and determination of clinical endpoints will be done as scheduled in table 1. All subjects will be managed to reach their glycemic, blood pressure and lipid goals according to guidelines. Subjects who discontinue study medication prematurely should continue to attend all subsequent study visits and be followed to the trial end date. The study plan of every visit is in Table 1.

Primary Objective: To determine if dapagliflozin + integrated CKD care program is more effective in reducing renal function progression than integrated CKD care program measured by Difference of eGFR slope after randomization

Secondary Objective: To determine if dapagliflozin + integrated CKD care program is more effective in reducing the composite of renal and cardiovascular endpoints than integrated CKD care program in a hierarchical testing sequence:

1. renal composite outcome: Cardiovascular or renal death, ESRD (sustained eGFR <5 mL/min/1.73m2, chronic dialysis or renal transplantation) and >50% sustained decline in eGFR (by the Modification of Diet in Renal Disease equation).
2. renal and heart failure outcome: renal composite outcome, acute kidney injury (increase in serum creatinine ≥1.5 times baseline within 7 days), and hospitalization for heart failure.
3. renal and cardiovascular outcome: renal and heart failure composite outcome and 5P-MACE (cardiovascular death, myocardial infarction, stroke, hospitalization for unstable angina or coronary/peripheral artery revascularization) Exploratory and biomarker objectives: as described in the protocol

Target subject population Briefly, subjects who are ≥20 years of age, eGFR ≥10 and ≤30 mL/min/1.73m2, eGFR decline >2.5 mL/min/1.73m2 in previous 12 months, and in in the pre-ESRD care and education program of Ministry of Health and Welfare of Taiwan for ≥1 months will be eligible for randomization.

Duration of treatment The anticipated duration of the study is at least 52 weeks. The study duration may be extended for further evaluation.

Investigational product, dosage and mode of administration Dapagliflozin 5-10 mg once daily (oral) + Integrated CKD Care program v.s. Integrated CKD Care program

Statistical methods Analysis sets: All patients randomized in the treatment period will be included in the intention-to-treat analysis for primary, secondary, and exploratory outcome irrespective of their protocol adherence and continued participation in the study. Per-protocol analysis will be on those that are 80% compliant. Because biomarkers may be done in a subset of patients, not all patients randomized will be included in the analysis for biomarker.

Sample size determination: The study aims to observe the differences of eGFR slope between 2 arms by 0.75 ml/min/1.73m2/yr to have 80% power accounting for the effect of treatment using a two-sided alpha of 5%. A total of approximately 120 subjects will be in the study group and 60 subjects will be in the control group based on the assumptions: (1) eGFR slope in control group: -5 ± 2.5 ml/min/1.73m2/yr, (2) Premature treatment discontinuation rate: 5% per year, (3) Overall lost-to-follow-up 1%, and (4) Duration of enrollment period: 52 weeks.

Primary efficacy analysis: A linear mixed effect model will be fitted to eGFR as a dependent variable for eGFR decline. The comparison of eGFR decline will be assessed by difference of eGFR decline between 2 arms from randomization to end of study.

Secondary efficacy analyses: In the analysis of the composite renal, renal and heart failure and renal and cardiovascular endpoints, dapagliflozin versus control will be compared using a Cox proportional hazards model with a factor for treatment group, stratified by randomization stratification factors (DM, baseline eGFR and baseline eGFR slope).

Exploratory objectives: In the analysis of the fluid overload and all hospitalization endpoints, dapagliflozin versus control will be compared using a Cox proportional hazards model with a factor for treatment group, stratified by randomization stratification factors (DM, baseline eGFR and baseline eGFR slope).

Safety analyses: Subjects in the safety analysis set will be included in the denominators for the summaries of adverse event, exposure, and concomitant medication data.

Multiplicity adjustment: A closed testing procedure will be implemented to control the overall type I error at 5% for a pre-specified hierarchical ordering of the primary and secondary endpoints.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of informed consent prior to any study specific procedures.
2. Aged ≥20 years at the time of consent.
3. eGFR ≥10 and ≤30 mL/min/1.73m2 (Modification of Diet in Renal Disease (MDRD) equation ) at randomization.
4. eGFR decline ≥2.5 mL/min/1.73m2 (≥ 3 measurements, simple linear regression) in one year before randomization.
5. In the pre-ESRD care and education program of Ministry of Health and Welfare of Taiwan (pre-ESRD program) for ≥3 months before randomization.

Exclusion Criteria:

1. Lupus nephritis, anti-neutrophil cytoplasmic autoantibody (ANCA)-associated vasculitis and organ transplantation.
2. Receiving therapy with an SGLT2 inhibitor within 8 weeks prior to enrolment or previous intolerance of an SGLT2 inhibitor.
3. Any condition outside the renal and CV disease area, with a life expectancy of less than 2 years based on investigator's clinical judgement.
4. Active malignancy requiring treatment at the time of visit 1.
5. Women of child-bearing potential who are not willing to use a medically accepted method of contraception throughout the study, OR women who have a positive pregnancy test at enrolment OR women who are breast-feeding.
6. Urinary tract obstruction (hydronephrosis, hydroureter and abnormal post-voiding residual urine volume under renal echography).
7. Frequent urosepsis (≥2 times in one year before enrollment) and history of Fournier's gangrene.
8. Inability of the patient, in the opinion of the investigator, to understand and/or comply with treatment, procedures and/or follow-up OR any conditions that, in the opinion of the investigator, may render the patient unable to complete the study.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2022-05-27 (Actual); Primary Completion 2024-08-31 (Actual); Study Completion 2024-08-31 (Actual)

PRIMARY OUTCOMES:
eGFR slope | from randomization to renal replacement therap, study completion or censoring event, upto 96 weeks
  eGFR decline after randomization between 2 arms

SECONDARY OUTCOMES:
Renal composite outcome | from randomization to study completion or censoring event, upto 96 weeks
  1. Cardiovascular or renal death.
  2. ESRD: sustained eGFR <5 mL/min/1.73m2, chronic dialysis or renal transplantation.
  3. >50% sustained decline in eGFR (by the Modification of Diet in Renal Disease equation).
Renal and heart failure composite outcome | from randomization to study completion or censoring event, upto 96 weeks
  1. renal composite outcome
  2. Acute kidney injury (increase in serum creatinine ≥1.5 times baseline within 7 days).
  3. Hospitalization for heart failure.
Renal and cardiovascular composite outcome | from randomization to study completion or censoring event, upto 96 weeks
  1. Renal and heart failure composite outcome.
  2. 5P-Major adverse cardiovascular events (cardiovascular death, myocardial infarction, stroke, hospitalization for unstable angina or coronary/peripheral artery revascularization).

CONTACTS AND LOCATIONS:
Overall Officials: Chi-Chih Hung, MD, Study Chair — Kaohsiung Medical University
Locations (1):
- Chi-Chih Hung, Kaohsiung City, Taiwan

IPD SHARING:
Plan to Share IPD: No
No plan.